CLINICAL TRIAL: NCT06504316
Title: A Multicenter, Randomized Control Clinical Trial on the Effect of Adsorptive Filter oXiris on Hemodynamics of Abdominal Septic Shock Patients
Brief Title: OXiris for Abdominal SEptic Shock (OASES Study)
Acronym: OASES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY2024-082-B
Record Dates: First submitted 2024-06-23; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock; Abdominal Sepsis; Multi Organ Failure; Blood Purification; AKI - Acute Kidney Injury
MeSH Terms: conditions — Shock, Septic; Intraabdominal Infections; Multiple Organ Failure; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Comparison two groups: intervention group (oXiris filter) and control group (ST 150 filter)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oXiris (Experimental): The subjects will be accepted oXiris filter at the first treatment session for 72 hours.
  Interventions: Device: CRRT filter
- ST 150 (Active Comparator): The subjects will be accepted ST 150 filter at the first treatment session for 72 hours.
  Interventions: Device: CRRT filter

INTERVENTIONS:
Device: CRRT filter — The subjects will be accepted CRRT using a filter for 72 hours. The subjects will be continued to CRRT or not after 72 hours (the first session of treatment) according to clinical situation by clinician decision. CRRT prescription: 1 Blood purification access: Central vein indwelling double lumen catheter (diameter 11F-13.5F) can be placed in femoral vein, internal jugular vein and subclavian vein; 2.Anti-coagulation prescription: Anticoagulant is used according clinical situation by clinician decision (such as heparin, sodium citrate, and so on); 3. Modality of CRRT: CVVH: blood flow 150-200ml/min; replacement fluid flow 30-35ml/kg/h (100% post-dilution).

SUMMARY:
This study innovatively utilizes multi-modal hemodynamic monitoring (Norepinephrine equivalence, NEE+Pulse indicator Continuous Cariac output, PiCCO) to investigate the optimal timing of initiation of oXiris in abdominal infection-associated septic shock patients and to investigate prognosis on sepsis phenotypes undergoing oXiris therapy.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction syndrome caused by dysregulated host responses to infection, which is one of the leading causes of death for critically ill patients and also a challenge for clinicians.

Abdominal infection is a common cause of septic shock, and is often transferred to intensive care unit (ICU) from emergency surgery, including appendectomy, cholecystectomy, intestinal repair or resection, incision and drainage of abscesses, and local debridement.

The oXiris (Baxter) hemofiltration membrane is the only one on the market with the ability to adsorb both cytokines and endotoxin. This, together with the renal replacement function and its antithrombogenic properties, makes it unique in that it brings together four important functions in a single device. Endotoxin adsorption occurs thanks to a significant number of positively charged free amino groups in Polyethylene imine (PEI), which bind to the negatively charged endotoxin. This capacity is much more important, as oXiris has significantly more PEI compared to previous membranes. Therefore, from the perspective of structural principle, oXiris is currently an ideal adsorptive blood purification filter, which can not only perform conventional renal replacement therapy, but also perform adsorptive therapy to provide extra-renal support for sepsis. Therefore, in terms of the structural properties of the membrane, oXiris is currently an ideal adsorptive blood purification filter for both conventional renal replacement therapy for renal dysfunction treatment and extra-renal support for sepsis with endotoxin adsorption therapy.

The investigaters hypothesis the adsorptive filter oXiris using for continuous renal replacement therapy (CRRT) can improve hemodynamic instability in abdominal septic shock patients, which rely on multimodal hemodynamics monitoring by PiCCO and ultrasound for early goal directed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Weight ≥30 kg;
3. Intra-abdominal infection (blood or abdominal drainage fluid culture positive for Gram-negative bacteria or suspected to be caused by a Gram-negative agent);
4. Diagnostic septic shock (Sepsis 3.0): Sepsis was defined as "life-threatening organ dysfunction caused by a dysregulated host response to infection" with organ dysfunction defined as an increase in qSOFA ⩾2 points. Septic shock was defined as sepsis requiring vasoactive therapy to maintain mean arterial pressure (MAP) ⩾ 65 mmHg and lactate elevation to >2 mmol/L despite adequate volume resuscitation;
5. The dose of norepinephrine⩾0.4ug/kg/min;
6. PCT⩾50ug/L, and/or IL-6⩾1000pg/ml;
7. AKI stage II/III (Kidney Disease Improving Global Outcomes, KDIGO grade);
8. Duration of septic shock ≤48 hours.

Exclusion Criteria:

1. Patients with highly contagious infectious diseases, such as tuberculosis;
2. Pregnant and lying-in woman or lactation period;
3. Infection of other sites (no abdominal infection like pneumonia, central nervous system infection and so on);
4. CRRT cannot be performed for various reasons;
5. Death is expected within 48 hours of admission to the ICU;
6. Previous renal replacement therapy;
7. Patients that underwent cardio-pulmonary resuscitation (CPR);
8. Patients who will not sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The dose of vasopressor agents | CRRT 0, 6, 12, 24, 48, 72 hours
  Decrease range of NEE after initiation of CRRT

SECONDARY OUTCOMES:
The value of PiCCO parameters | CRRT 0, 6, 12, 24, 36, 48, 72 hours
  Increase range of cardiac index (CI) and systemic vascular resistance index (SVRI) after initiation of CRRT
The level of inflammatory markers | CRRT 0, 12, 24, 48, 72 hours
  Decrease range of serum procalcitonin (PCT), interleukin-6 (IL-6) level after initiation of CRRT
The severity of illness score Severity of illness score | CRRT 0, 24, 48, 72 hours
  Decrease range of Acute Physiology and Chronic Health Evaluation II (APACHE II) and Sequential Organ Failure Assessment (SOFA) score during the first 72 hours
The time of hospital stay | From date of randomization until the date of end of followup
  Length of hospital and ICU stay
The number of subjects of survival and kidney recovery | Day 28, 60, 90
  Survival and kidney recovery

OTHER OUTCOMES:
The nmber of subjects of survival in phenotypes of septic shock | Day 28, 60, 90
  The survival of various phenotypes of septic shock
Filter lifespan | From time of filter initiation using until the time of filter changed or CRRT stop (if filter no changed)
  Duration of oXiris filter using and timing of changing filter

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

REFERENCES:
- [Derived] Chen J, Zhang Z, Gao J, Liu Y, Zhu B, Gao Y, Zhuang Y, Zhu M. A multicentre, randomised controlled clinical trial evaluating the effect of the adsorptive filter oXiris on haemodynamics in abdominal septic shock patients requiring continuous renal replacement therapy (Oxiris for Abdominal SEptic Shock study). BMJ Open. 2025 Jul 8;15(7):e094792. doi: 10.1136/bmjopen-2024-094792. PMID 40633959